CLINICAL TRIAL: NCT00663650
Title: A Randomized Clinical Trial in the Surgical Treatment of Basal Cell Carcinoma of the Eyelid: Surgical Excision With Frozen Section vs. Permanent Section Control
Brief Title: Periocular Basal Cell Carcinoma (BCC): Permanent vs. Frozen Section Pathological Control
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Responsible Party: Vladimir Kratky, MD, FRCSC, Department of Ophthalmology, Queen's University, Kingston, ON, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal Cell Carcinoma; BCC; Periocular BCC; Frozen Section Control; Permanent Section Control; Recurrence Rates
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Permanent Section Control
  Interventions: Procedure: Permanent Section Control
- 2 (Active Comparator): Frozen Section Control
  Interventions: Procedure: Frozen Section Control

INTERVENTIONS:
Procedure: Permanent Section Control — After surgical excision of the tumor, margins will be sent for permanent section pathologic control to determine if the tumor was completely excised
  Arms: 1
Procedure: Frozen Section Control — After surgical excision of the tumor, tumor edges will be analyzed by frozen section at the time of surgery. If tumor margins are positive with the frozen section, additional tissue will be excised and analyzed again. This process will be repeated until all tissue edges are clear of tumor. Finally, the area of tumor excision will be surgically reconstructed.
  Arms: 2

SUMMARY:
This study is an equivalency study designed as a randomized clinical trial. Patients with a biopsy proven nodular periocular basal cell carcinoma (BCC) who have agreed to have surgical excision will be eligible. Study patients will undergo surgical excision of the lesion and then be randomized to having frozen section or permanent section pathological control. For those patients randomized to permanent section control the sample will be sent to pathology and surgical reconstruction will be performed. Patients randomized to frozen section will have additional margins re-excised before reconstruction depending on the pathologic results. Tumor clearance rates after surgical excision will be compared between the two techniques as a primary study question. Patients will be followed long-term to determine recurrence rates in the two groups. The study is designed to determine if the two techniques are equivalent within a given margin of error with respect to outcome measures.

DETAILED DESCRIPTION:
Basal cell carcinoma (BCC) accounts for 80-90% of skin cancers and is the most common skin cancer of the periocular region. Surgical excision is considered the gold-standard in therapy. Previous literature has shown comparable recurrence rates of BCC between surgical excision with frozen section control and surgical excision and permanent section control. To data, there are no prospective studies comparing frozen section control with permanent section control. We hypothesize that short term tumor clearance rates between frozen section and permanent section control will be similar and that long-term tumor recurrence rates will be similar between the two techniques. If we find that these two treatment options are equivalent with respect to margin control and recurrence rates, then considerable time and money savings can be accrued through using permanent section control amongst patients with periocular BCC.

The study design is a single-blind randomized controlled trial. Patients who have already agreed to surgical excision of nodular type periocular BCC will be eligible. All patients will undergo a detailed informed consent process. All patients will undergo a punch biopsy to confirm the histopathological diagnosis of BCC. The study design will be a single-blinded, randomized clinical trial. Statistically, the study will be designed as an equivalency study. Prior to randomization the BCC will be excised with 3mm clinical margins in a standard fashion. Subjects will then be randomized to one of two groups: 1. Frozen section control; 2. Permanent section control. For those patients randomized to permanent section control the clinical sample will be sent for pathologic analysis and surgical reconstruction will be performed immediately using standard oculoplastic techniques. Patients randomized to frozen section will have additional margins re-excised if necessary depending on the pathologic results. Oculoplastic reconstruction will be performed after all margins are clear. Patients will undergo examinations at the following times to assess for clinical recurrence: 1. 2 weeks and as necessary thereafter to assess surgical result and wound healing, 2. 6 months, 3. 1 year, 4. yearly up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or greater
* Diagnosed with clinically nodular BCC in the periocular region confirmed by tissue biopsy
* Agreeable and medically able to undergo surgical excision of the BCC
* Able to give informed consent and consent has been signed
* Able to return for all follow up visits

Exclusion Criteria:

* BCC greater than 2cm in diameter (based on clinical examination)
* Patient with a medical condition predisposing to multiple BCC's (ex. basal cell nevus syndrome)
* Recurrent BCC's (i.e. a BCC that has been treated previously by surgical or other modality and has recurred will not be eligible)
* Clinically aggressive morpheaform subtype of BCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2008-08; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of BCC's that are pathologically clear of tumor cells in the permanent section group compared with the frozen section group (presumably clear for all patients). | 1.5 years

SECONDARY OUTCOMES:
Clinical recurrence at 3 years | 4.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Kratky, MD, FRCSC, Principal Investigator — Department of Ophthalmology, Queen's University, Kingston, ON
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada